CLINICAL TRIAL: NCT03817801
Title: Comparison of Scoring Balloon and Conventional Balloon Predilation Before Drug Coated Balloon for de Novo Lesion in Patients With High Bleeding Risk: A Randomized, Single-center, Pilot Study
Brief Title: Comparison of Scoring Balloon and Conventional Balloon Predilation Before Drug Coated Balloon for de Novo Lesion in Patients With High Bleeding Risk
Acronym: PREPARE-NSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Junjie Zhang, Vice Director of Cardiovascular Department, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFH20190104
Record Dates: First submitted 2019-01-21; First posted 2019-01-28 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will undergo 1:1 randomization to either non-slip element (NSE) predilation which will be the treatment group or non-compliant (NC) balloon predilation which will be the control group. The initiation of the trial is defined as the time of randomization. After study subjects' enrollment and randomization, the study intervention will take place immediately. The follow-up visits for the primary endpoint are scheduled at 1and 6 months after the index procedure.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will remain blinded until the final study results are released.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-slip element (NSE) predilation (Experimental): In the NSE predilation group, NSE predilation will be performed for all lesions preparation before drug-coated balloon (DCB) treatment.
  Interventions: Device: NSE balloon
- non-compliant (NC) balloon predilation (Active Comparator): In the NC balloon predilation group, NC balloon predilation will be performed for all lesions preparation before DCB treatment.
  Interventions: Device: NC balloon

INTERVENTIONS:
Device: NSE balloon — NSE (Goodman®) predilation + DCB (Sequent® Please) treatment
  Arms: non-slip element (NSE) predilation
Device: NC balloon — NC balloon predilation + DCB (Sequent® Please) treatment
  Arms: non-compliant (NC) balloon predilation

SUMMARY:
This study is designed to investigate whether scoring balloon (non-slip element, NSE) predilation compared to non-compliant (NC) balloon predilation for de novo lesion in patients with high bleeding risk and planning to receive drug-coated balloon (DCB) treatment will lead to lower change in minimal lumen area (MLA) at 6 months by intravascular ultrasound (IVUS).

DETAILED DESCRIPTION:
This is a pilot study that aim to enroll 60 subjects with high bleeding risk.

All patients with coronary artery stenosis suitable for DCB treatment will undergo 1:1 randomization either to NSE predilation or NC balloon predilation using a randomization schedule.

All subjects will be screened according to the predefined inclusion and exclusion criteria per protocol and will further undergo IVUS before DCB treatment. Data and images will be collected during the index procedure, and at the predefined 6-month IVUS follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* De Novo lesion, suitable for intravascular ultrasound (IVUS) and fractional flow reserve (FFR) test;
* Coronary artery disease (CAD) patients with high risk of bleeding

Exclusion Criteria:

* Previous coronary artery bypass graft (CABG) patients
* Stent implantation in the target vessel
* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2
* Acute ST segment elevation myocardial infarction (STEMI) within 48 hours
* Contraindications to contrast media, antiplatelet therapy, or paclitaxel
* Cardiac shock
* Pregnancy
* Expected life less than 12 months

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The absolute change in minimal lumen area (MLA) | 6 months
  The absolute change in MLA from post-procedure to 6-month follow-up identified by intravascular ultrasound (IVUS)

SECONDARY OUTCOMES:
Bailout drug-eluting stents (DES) implantation rate | During procedure
  Bailout DES implantation rate during procedure by angiographic criteria
Fractional Flow Reserve (FFR) value | immediately after balloon predilation
  FFR value after balloon predilation measured by FFR
Minimum lumen area (MLA) | immediately after procedure
  MLA after procedure by IVUS
Minimum lumen diameter (MLD) | immediately after procedure
  MLD after procedure by IVUS
Plaque burden | immediately after procedure
  Plaque burden after procedure by IVUS
Dissection | immediately after procedure
  Dissection after procedure by IVUS
Atheroma volume | immediately after procedure
  Atheroma volume after procedure by IVUS
The diameter stenosis of target lesion | 6 months
  The diameter stenosis of target lesion from post-procedure to 6-month follow-up by angiography
The late lumen loss of target lesion | 6 months
  The late lumen loss of target lesion from post-procedure to 6-month follow-up by angiography
The binary restenosis of target lesion | 6 months
  The binary restenosis of target lesion from post-procedure to 6-month follow-up by angiography
The composite of cardiac death, myocardial infarction, target lesion revascularization (TLR), and target lesion thrombosis | 6 months
  The composite of cardiac death, myocardial infarction, TLR, and target lesion thrombosis at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No